CLINICAL TRIAL: NCT05732740
Title: Evaluating the Feasibility and Preliminary Effect of Empower@Home: Connected for Depression, Social Isolation, and Loneliness Among Older Adults.
Brief Title: Empower@Home:Connected - Feasibility and Preliminary Effect Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Xiaoling Xiang, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00212950-Group
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Depression; Loneliness; Social Isolation; Depressive Disorder; Mood Disorders; Mental Disorder
MeSH Terms: conditions — Depression; Social Isolation; Depressive Disorder; Mood Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: The purpose of this research project is to assess the preliminary effect of a novel internet-based cognitive behavioral therapy (iCBT) program called Empower@Home:Connected. The program is delivered in small groups remotely. It is intended to decrease depression, social isolation, and loneliness in participants by encouraging participants to take part in meaningful and enjoyable activities while challenging problematic thinking patterns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants will participant in 9 weekly group-based sessions
  Interventions: Behavioral: Empower@Home:Connected

INTERVENTIONS:
Behavioral: Empower@Home:Connected — Cognitive behavioral therapy

SUMMARY:
This single-group trial will evaluate the feasibility and preliminary effect of a novel group-based cognitive behavioral therapy program for older adults with elevated depressive symptoms. Participants will complete the program remotely in small groups.

DETAILED DESCRIPTION:
Depression affects up to 40% of homebound seniors, but most do not receive psychotherapy due to various access barriers. This study focuses on developing community-based solutions to reduce access barriers. In a previously approved project HUM00207612, the investigators tested the feasibility of a novel internet-based cognitive behavioral therapy (iCBT) program called Empower@Home. This study will test an adapted version of Empower@Home called Empower@Home: Connected that is delivered in a group format and also addresses social isolation and loneliness. Recruitment methods include 1) referrals from social service agencies, 2) advertisements on social media, local news outlets, and the program website, and 3) research participant registries.

The intervention involves attending 9 group sessions. The sessions are facilitated by a mental health professional and involve psychoeducational material, cognitive-behavioral therapy exercises, and socialization. Sessions will occur on 9 consecutive weeks and will last approximately 90 minutes. Participants will complete a comprehensive baseline assessment and post-test. Each assessment will take between 40-60 minutes to complete over the phone. Recruitment will occur between January and April 2023, 20-25 participants will be recruited. All participants will receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* >=60 years
* have at least mild depressive symptoms, based on PHQ-9 >=8
* are willing to participate

Exclusion Criteria:

* Probable cognitive impairment based on the Blessed Orientation, Memory, and Concentration scale (score >9).
* They do not speak English
* have active suicidal ideation, defined as moderate to high risk based on the 6-item Columbia-Suicide Severity Rating Scale (C-SSRS)
* Have a terminal illness or unstable physical health with a high risk of hospitalization within the next 3 months
* Have severe vision impairment that can not be corrected
* Have probable substance use disorders as assessed by the 4-item CAGE screener (>=2 on the CAGE AND have not been sober for at least one year)
* Have a self-reported psychotic disorder or bipolar disorder

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 | Change from baseline PHQ9 to post-test at 9 weeks
  Changes in 9-item standardized measure of depression symptom severity. PHQ-9 scores range from 0 to 27, with higher scores indicating more depressive symptoms.
Changes in De Jong Gierveld Scale | Change from baseline De Jong Gierveld Scale to post-test at 9 weeks
  Change in 6-item De Jong Gierveld Short Scale for Emotional and Social Loneliness. Scores range from 0 to 6, with higher scores indicating more loneliness.
Changes in Patient-Reported Outcomes Measurment Information Systems - Social Isolation. | Change from baseline PROMIS-Social Isolation to post-test at 9 weeks
  Changes in 8-item Patient-Reported Outcomes Measurment Information Systems - Social Isolation. PROMIS - SI scores range from 0 to 32, with higher scores indicating higher social isolation.

SECONDARY OUTCOMES:
Changes in Generalized Anxiety Disorder Assessment-7 | Change inGeneralized Anxiety Disorder Assessment-7 baseline to post-test at 9 weeks
  Changes in 7-item standardized measure for severity of anxiety symptoms. GAD-7 Scores range from 0 to 21, with higher values indicating higher anxiety.
Changes in Health Related Quality of Life | Change from baseline Health-Related Quality of Life to post-test at 9 weeks
  Change in 5-item Health-Related Quality of Life. EQ5D-5L Scores range from 0 to 20 with higher scores indicating lower health related quality of life.
Changes in Patient-Reported Outcomes Measurment Information Systems- Global Health | Change from baseline PROMIS-Global Health to post-test at 9 weeks
  Change in 9-item Patient-Reported Outcomes Measurment Information Systems - Global Health. PROMIS-GH scores range from 9 to 45, with higher scores meaning poorer global health..

CONTACTS AND LOCATIONS:
Overall Officials: Jay Kayser, MSW, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No